CLINICAL TRIAL: NCT00674193
Title: A Pharmacokinetic-Pharmacodynamic-Pharmacogenetic Study of Actinomycin-D and Vincristine in Children With Cancer
Brief Title: Evaluating Dactinomycin and Vincristine in Young Patients With Cancer
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ADVL06B1; NCI-2009-00362 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL06B1 (Other: Children's Oncology Group); CDR0000559243 (Other: Clinical Trials.gov); U10CA098543 (NIH)
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Childhood Acute Lymphoblastic Leukemia; Childhood Rhabdomyosarcoma; Childhood Soft Tissue Sarcoma; Ewing Sarcoma; Ewing Sarcoma of Bone; Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor (PNET); Unspecified Childhood Solid Tumor, Protocol Specific; Wilms Tumor and Other Childhood Kidney Tumors
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Sarcoma, Ewing; Neuroectodermal Tumors, Primitive, Peripheral; Wilms Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational (pharmacological study): Patients undergo blood and urine collection prior to, periodically during, and after treatment with dactinomycin and vincristine for pharmacokinetic, pharmacodynamic, and pharmacogenetic analysis. Samples are analyzed using a liquid chromatography-tandem mass spectrometry assay. Genomic DNA extracted from peripheral blood mononuclear cells is isolated and analyzed by polymerase chain reaction and genotyping assays for genetic variation in genes relevant to the pharmacology of dactinomycin and vincristine.
  Interventions: Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This laboratory study is evaluating how well dactinomycin and vincristine work in treating young patients with cancer. Studying samples of blood and urine in the laboratory from patients with cancer may help doctors learn how dactinomycin and vincristine affect the body and how patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the pharmacokinetics (PKs) of dactinomycin in infants, children, and adolescents with cancer.

II. To identify demographic or physiological factors that are determinants of dactinomycin disposition.

III. To characterize the PKs of vincristine (VCR) in infants, children, and adolescents with cancer.

IV. To identify demographic or physiological factors that are determinants of VCR disposition.

SECONDARY OBJECTIVES:

I. To examine the correlation of dactinomycin and VCR systemic exposure metrics with toxicity outcomes.

II. To explore the PK, pharmacodynamic, and pharmacogenetic relationships of dactinomycin and VCR in children with cancer.

OUTLINE: This is a multicenter study.

Patients undergo blood and urine collection prior to, periodically during, and after treatment with dactinomycin and vincristine for pharmacokinetic, pharmacodynamic, and pharmacogenetic analysis. Samples are analyzed using a liquid chromatography-tandem mass spectrometry assay. Genomic DNA extracted from peripheral blood mononuclear cells is isolated and analyzed by polymerase chain reaction and genotyping assays for genetic variation in genes relevant to the pharmacology of dactinomycin and vincristine.

After the final pharmacokinetic sample is collected, patients are followed for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer, including, but not limited to, any of the following:

  * Acute lymphoblastic leukemia
  * Ewing sarcoma
  * Rhabdomyosarcoma
  * Soft tissue sarcoma
  * Wilms tumor
* Due to receive or receiving dactinomycin and/or vincristine as a component of cancer treatment on another clinical trial
* Able to comply with study requirements
* Other concurrent chemotherapeutic agents allowed

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with a diagnosis of cancer, including, but not limited to, any of the following: Acute lymphoblastic leukemia, Ewing sarcoma, Rhabdomyosarcoma, Soft tissue sarcoma, Wilms tumor who are due to receive or receiving dactinomycin and/or vincristine as a component of cancer treatment on another clinical trial
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2008-02; Primary Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Population PK parameters for dactinomycin and VCR | Not Provided
Demographic and/or physiological factors that are determinants of dactinomycin and VCR disposition | Not Provided

SECONDARY OUTCOMES:
Pharmacokinetic (PK), pharmacodynamic (PD), and pharmacogenetic characteristics of dactinomycin and vincristine (VCR) | Not Provided
Pharmacogenetic profiles of patients receiving dactinomycin and VCR | Not Provided
Correlation between genetic variation in drug metabolizing enzymes and drug transporters and observed drug PKs and PDs in children | Not Provided
Creation of population PK and PD models to assess the effect of drug exposure on toxicity and outcomes | Not Provided
Correlation of dactinomycin and VCR systemic exposure metrics with toxicity outcomes | Not Provided

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, Principal Investigator — Children's Oncology Group
Locations (38):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Childrens Hospital of Orange County, Orange, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - Nemours Childrens Clinic - Orlando, Orlando, Florida
  - Saint Joseph Children's Hospital of Tampa, Tampa, Florida
  - University of Illinois, Chicago, Illinois
  - Childrens Memorial Hospital, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Mission Hospitals Inc, Asheville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Hospital Sainte-Justine, Montreal, Quebec, Canada